CLINICAL TRIAL: NCT05495568
Title: A Randomized, Active-Controlled, Double-Blind, Phase 3 Study to Compare Pharmacokinetics, Efficacy, and Safety of CT-P17 With Humira in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: To Compare Pharmacokinetics, Efficacy, and Safety of CT-P17 With Humira in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P17 3.3; 2022-002336-31 (EudraCT Number)
Record Dates: First submitted 2022-08-07; First posted 2022-08-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
MeSH Terms: interventions — CT-P17

STUDY DESIGN:
Intervention Model Description: Interchangeability study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switching CT-P17 (Experimental): On Day 1, Week 0, patients will be enrolled in the study and receive Humira. The patients will receive initial dose of Humira (80 mg; 2 shots of 40 mg) on Day 1 and Humira (40 mg) EOW starting one week after the initial dose until Week 11.
  Prior to the study drug administration at Week 13, patients will be randomized to receive either CT-P17 (40 mg) or Humira (40 mg) and the CT-P17 Switching group will receive CT-P17 (40mg) at Week 13, Week 15, Week 21, Week 23 and Week 25. The Switching group will receive Humira at Week 17 and Week 19.
  From Week 27, patients will receiAve CT-P17 (40 mg) EOW only as open-label up to Week 49.
  Interventions: Biological: CT-P17; Biological: EU-approved Humira
- Humira maintenance (Active Comparator): On Day 1, Week 0, patients will be enrolled in the study and receive Humira. The patients will receive initial dose of Humira (80 mg; 2 shots of 40 mg) on Day 1 and Humira (40 mg) EOW starting one week after the initial dose until Week 11.
  Prior to the study drug administration at Week 13, patients will be randomized to receive either CT-P17 (40 mg) or Humira (40 mg) and the Humira maintenance group will receive Humira (40mg) EOW up to Week 25.
  From Week 27, patients will receive CT-P17 (40 mg) EOW only as open-label up to Week 49.
  Interventions: Biological: CT-P17; Biological: EU-approved Humira

INTERVENTIONS:
Biological: CT-P17 — CT-P17 40mg will be subcutaneous administered
Biological: EU-approved Humira — subcutaneous administration

SUMMARY:
This is a Phase 3 Study to Compare Pharmacokinetics, Efficacy and Safety of CT-P17 with Humira in Patients with Moderate to Severe Chronic Plaque Psoriasis

DETAILED DESCRIPTION:
CT-P17 is a recombinant human monoclonal antibody containing the active ingredient adalimumab (human TNF-α blocker). CT-P17 is a drug product being developed by CELLTRION, Inc. and being compared to both the EU-approved Humira® and US-licensed Humira®. In this study, Pharmacokinetics, Efficacy and Safety of CT-P17 will be evaluated in patients with Moderate to Severe Chronic Plaque Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged 18 to 75 years old, both inclusive.
2. Patient has had a diagnosis of chronic plaque psoriasis for at least 24 weeks prior to the first administration of the study drug (Day 1).
3. Patient has stable moderate to severe plaque psoriasis with or without psoriatic arthritis at both Screening and at the time of the first administration of the study drug (Day 1) as defined by:

   * Psoriasis Area and Severity Index (PASI) score of 12 or greater and
   * Static Physician's Global Assessment (sPGA) score of 3 or greater and
   * Body Surface Area (BSA) affected by plaque psoriasis of 10% or greater.
4. Patient who is a candidate for systemic therapy or phototherapy.
5. Patient (or legal guardian, if applicable) is informed of the full nature and purpose of the study, including possible risks and side effects, is able to cooperate with the investigator and is given ample time and opportunity to read and understand verbal and/or written instructions, and signs the written informed consent form with date prior to participation in the study.
6. Female patient who is considered of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree to use highly effective methods of contraception consistent with local regulations during the course of the study and at least 20 weeks following discontinuation of study drug (excluding women who are not of childbearing potential). Examples include the following:

   1. Combined (estrogen and progestogen containing) or progestogen-only hormonal contraceptives associated with inhibition of ovulation
   2. Intrauterine device or intrauterine hormone-releasing system
   3. True abstinence, when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to investigational drug, and withdrawal are not acceptable methods of contraception.

Male patient who is sexually active with a woman of childbearing potential must agree to use the highly effective method described as above or medically acceptable methods of contraception (e.g., male or female condom AND additional hormonal or barrier method by female partner) consistent with local regulations during the study and for 20 weeks following discontinuation of study drug. If patient or their partner has been surgically sterilized for less than 24 weeks prior to the date of informed consent form (ICF), they also must agree to use method(s) of contraception as described above. Postmenopausal female patients must have experienced their last menses more than 1 year prior to the date of ICF without an alternative medical cause to be classified as not of childbearing potential.

Exclusion Criteria:

1. Patient diagnosed with forms of psoriasis other than chronic plaque (e.g., pustular, erythrodermic or guttate psoriasis) or medication-induced psoriasis (e.g., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium).
2. Patient who has previously received investigational or licensed product of tumor necrosis factor (TNF) α inhibitor for any purposes.
3. Patient who has prior exposure to 2 or more biologic agents considered by the investigator to affect the outcome of the study. Patient with 1 prior biologic agent which is not classified as TNF-α inhibitor (e.g., interleukin [IL]-17, IL-12/23, IL-23 blocker) can be enrolled after 5 half-lives prior to the first administration of the study drug (Day 1).
4. Patient who has allergies to any of the excipients of study drug or materials of device or any other murine and human proteins, or patient with a hypersensitivity to immunoglobulin products.
5. Patient who currently has, or has a history of, any of the following infections:

   1. A known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C (active or carrier state) or syphilis. However, a patient with past hepatitis B virus and/or hepatitis C virus is allowed if resolved.
   2. Recurrent herpes zoster or other chronic or recurrent infection within 6 weeks prior to the first administration of the study drug (Day 1).
   3. Past or current granulomatous infections or other severe or chronic infections (such as sepsis, abscess, opportunistic infections, or invasive fungal infections such as histoplasmosis). A patient who has a past diagnosis with sufficient documentation of complete resolution of the infection can be enrolled in the study.
   4. Acute infection requiring oral antibiotics within 2 weeks prior to the first administration of the study drug (Day 1) or a serious infection associated with hospitalization and/or which required parenteral injection of antibiotics within 24 weeks before Day 1.
6. Patient who currently has, or has a history of, any of the following TB conditions:

   1. Patient who has a history of TB or a current diagnosis of TB. A patient who has a previous diagnosis of active TB cannot be enrolled in the study even if there is sufficient documentation of complete resolution of active TB.
   2. Patient who has had exposure to a person with active TB such as first-degree family members or co-workers.
   3. Patient who has an indeterminate result for interferon-γ release assay (IGRA) or latent TB (defined as a positive result of IGRA with a negative examination of chest X-ray) at Screening. A patient who has a previous diagnosis of latent TB cannot be enrolled despite sufficient documentation of prophylaxis. If the result of the IGRA is indeterminate at Screening, 1 retest will be possible during the Screening period. If the repeated IGRA result is indeterminate again or positive, the patient will be excluded from the study. If the repeated IGRA result is negative, the patient can be enrolled in the study.
7. Patient who has a medical condition including one or more of the following:

   1. Classified as Class III obesity by WHO classification (body mass index≥40 kg/m2)
   2. Diabetes mellitus considered by the investigator to be clinically significant and uncontrolled, even after insulin treatment.
   3. Uncontrolled hypertension (as defined by systolic blood pressure [BP] ≥160 mmHg or diastolic BP ≥100 mmHg).
   4. Active ongoing inflammatory or autoimmune disease other than chronic plaque psoriasis and psoriatic arthritis, that may confound the evaluation of the effect of the study drug.
   5. History of a known malignancy within the previous 5 years prior to the first administration of the study drug (Day 1) except completely excised and cured squamous carcinoma of the uterine cervix in situ, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma.
   6. New York Heart Association class III or IV heart failure, severe uncontrolled cardiac disease (unstable angina or clinically significant electrocardiogram [ECG] abnormalities), or myocardial infarction within 24 weeks prior to the first administration of the study drug (Day 1).
   7. History of organ transplantation, including corneal graft/transplantation.
   8. Any underlying condition (e.g., metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) that, in the opinion of the investigator significantly immunocompromises the patient and/or places the patient at unacceptable risk for receiving an immunomodulatory therapy.
   9. Pre-existing or recent-onset central or peripheral nervous system demyelinating disease, including multiple sclerosis, optic neuritis and Guillain-Barre syndrome.
   10. Any other serious acute or chronic medical or psychiatric condition that could increase the risk associated with study participation or study drug administration or that could interfere with the interpretation of study results.
   11. History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion.
8. Patient who has the following laboratory abnormalities:

   1. Hemoglobin ≤8.0 g/dL (SI [Système International d'Unités] units: ≤80 g/L or 4.96 mmol/L).
   2. Platelet count <75× 103 cells/µL (SI units: <75 × 109 cells/L).
   3. Absolute neutrophil count <1.5 × 103 cells/µL (SI units: <1.5 × 109 cells/L).
   4. Alanine aminotransferase or aspartate aminotransferase >3.0 × upper limit of normal (ULN).
   5. Serum creatinine >1.5 × ULN or an estimated creatinine clearance level ≤50 mL/min (by Cockcroft-Gault formula) (SI units: 0.84 mL/s).
9. Patient who has received or plans to receive any of following prohibited medications or treatments:

   1. Topical treatment for psoriasis or any other skin condition (e.g., corticosteroids, vitamin D analogues, pimecrolimus, retinoids, salicylvaseline, salicylic acid, lactic acid, tacrolimus, tar, urea, α-hydroxy or fruit acids) within 2 weeks prior to the first administration of the study drug (Day 1). However, low-potency topical corticosteroids (Class 6 or 7) applied to the face and intertriginous areas are permitted during study participation to reduce patient's burden with a restriction of use within 12 hours prior to study visits requiring PASI or sPGA measures. Bland moisturizers/emollients not containing pharmacological active ingredients are permitted for treatment of psoriasis during study participation, but these should not be used within 12 hours before study visits when efficacy assessments are going to be performed.
   2. Ultraviolet A or B phototherapy (without oral psoralen) or psoralen with Ultraviolet A photochemotherapy for the treatment of psoriasis within 4 weeks prior to the first administration of the study drug (Day 1).
   3. Any systemic immunomodulating treatments (e.g., MTX, cyclosporine A, corticosteroids, cyclophosphamide, and other systemic nonbiologic therapies [e.g., apremilast, tofacitinib]) within 4 weeks prior to the first administration of the study drug (Day 1).
   4. Any other investigational device or medical product within 4 weeks prior to the first administration of the study drug (Day 1) or 5 half-lives, whichever is longer.
   5. Initiation or dose modification of drugs that may aggravate psoriasis (e.g., beta-blockers, calcium channel blocker or lithium) within 4 weeks prior to the first administration of the study drug (Day 1). Patients who have been on stable dose without exacerbation of psoriasis for at least 4 weeks prior to the first administration of the study drug (Day 1) can be enrolled, however, the same dose should remain throughout the study.
10. Patient who has received live or live-attenuated vaccine within 4 weeks prior to the first administration of the study drug (Day 1), or any planned live or live-attenuated vaccination during the study period.
11. Herbal remedies that could affect the outcome of the study within 2 weeks prior to the first administration of the study drug (Day 1).
12. Patient not willing to limit UV light exposure (e.g., sunbathing and/or the use of tanning devices) during the course of the study.
13. Patient with inability or unwillingness to undergo repeated venipuncture (e.g., because of poor tolerability or lack of access to veins).
14. Female patient who is currently pregnant or breastfeeding, or plans to become pregnant or breastfeed within 20 weeks of the last dose of study drug. Male patient who is planning to donate sperm or father a child within 20 weeks of the last dose of study drug.
15. Patient who currently abuses alcohol or drugs or has a history of alcohol or drug abuse within 1 year from Screening.
16. Patient is vulnerable (e.g., employees of the study center or any other individuals involved with the conduct of the study, or immediate family members of such individuals, persons kept in prison, or other institutionalized persons by law enforcement).
17. Patient who, in the opinion of their physician or the investigator, should not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate the pharmacokinetics (PK) similarity between patients receiving Humira continuously and those who alternate between Humira and CT-P17 in terms of Area under the concentration-time curve over the dosing interval (AUCtau, 25-27) | Week 25-27
To demonstrate the pharmacokinetics (PK) similarity between patients receiving Humira continuously and those who alternate between Humira and CT-P17 in terms of Maximum serum concentration during the dosing interval (Cmax, 25-27) | Week 25-27

SECONDARY OUTCOMES:
To evaluate Pharmacokinetics (PK) Pharmacokinetics (PK) parameter: Time to maximum serum concentration during the dosing interval (Tmax, 25-27) | Week 25-27
To evaluate Pharmacokinetics (PK) Pharmacokinetics (PK) parameter: Trough concentration (Ctrough) | up to Week 52
To evaluate Efficacy: Mean % improvement from baseline in PASI (Psoriasis Area Severity Index) score | up to Week 52
To evaluate Efficacy: Proportion of patients achieving at least 50/75/90/100% improvement from baseline in PASI (PASI 50/75/90/100) | up to Week 52
To evaluate Efficacy: Proportion of patients with an sPGA (Static Physician's Global Assessment) score on a 5-point scale of clear (0) or almost clear (1) | up to Week 52
To evaluate Safety: AEs (including serious AEs) by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | up to Week 52
To evaluate Safety: AEs of special interest by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | up to Week 52
To evaluate Safety: Immunogenicity of Switching and Humira maintenance will be assessed by anti-drug antibody and neutralizing antibody test in validated immunoassay. | up to Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- CT-P17 3.3 investigational site, Tallinn, Estonia

REFERENCES:
- [Derived] Pariser DM, Lebwohl MG, Jaworski J, Trefler J, Daniluk S, Dudek A, Baran W, Owczarek W, Brzewski P, Sikora M, Krogulec M, Kim S, Suh J, Choi E, Cha J, Lee H, Lee S, Koo JY. CT-P17 Adalimumab Biosimilar in Patients with Moderate-to-Severe Chronic Plaque Psoriasis: An Open-Label Extension of a Phase 3 Interchangeability Study. Dermatol Ther (Heidelb). 2025 May;15(5):1079-1092. doi: 10.1007/s13555-025-01383-5. Epub 2025 Mar 27. PMID 40148673
- [Derived] Lebwohl MG, Koo JY, Jaworski J, Trefler J, Daniluk S, Dudek A, Baran W, Owczarek W, Kolinek J, Brzewski P, Sikora M, Krogulec M, Kim S, Bae Y, Jeon D, Choi E, Cha J, Lee H, Choi S, Pariser DM. Repeated Switching Between CT-P17 and EU Reference Adalimumab in Patients with Moderate-to-Severe Chronic Plaque Psoriasis: A Randomized, Double-Blind, Active-Controlled, Phase 3, Interchangeability Study. Adv Ther. 2025 Mar;42(3):1582-1599. doi: 10.1007/s12325-024-03100-8. Epub 2025 Feb 11. PMID 39932677